CLINICAL TRIAL: NCT03597776
Title: Intravenous Lidocaine in Total Knee Replacement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chi-Wai Cheung, Clinical Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW18-276
Record Dates: First submitted 2018-07-15; First posted 2018-07-24 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Acute Pain
Keywords: intravenous lidocaine; pain; total knee replacement; spinal anaesthesia
MeSH Terms: conditions — Acute Pain; Pain | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine Group (Experimental): Bolus of intravenous lidocaine of 2mg/kg over 5 mins will be given before skin incision.
  Interventions: Drug: Lidocaine
- Placebo Group (Placebo Comparator): Normal Saline of 2mg/kg over 5 mins will be given as bolus before skin incision
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Lidocaine — Bolus of lidocaine will be given over 5 minutes before skin incision
  Other Names: Lignocaine HCL inj 2% B.P.
  Arms: Lidocaine Group
Drug: Saline — Bolus of saline will be given over 5 minutes before skin incision
  Arms: Placebo Group

SUMMARY:
Osteoarthritis of knees and hips is a common medical problem present in elderly, which poses signiﬁcant impairment to their mobility, independence, and quality of life. Despite the availability of conservative treatment, such as simple analgesics and physiotherapy, total joint replacement is the only curative option for this disease entity.

The latter, however, is not without risk. A study by Poulakka has demonstrated that patients with poor pain control in the postoperative period were three to ten times more likely to develop chronic pain, which may signiﬁcantly impair the patients' functional status and quality of life.

Optimal pain control is therefore essential in facilitating rehabilitation and in preventing long-term morbidities.

Lidocaine [2-(diethylamino)-N-(2,6-dimethylphenyl)acetamide] is an amide local anaesthetic that is characteristically fast in onset and short in duration of action. As such, it has long been used for providing regional anaesthesia for operation, but with limited role in terms of post operative analgesia.

Recently, intravenous infusion of lidocaine has been shown to be safe and eﬀective in reducing post operative pain (resting and dynamic), opioid consumption, and chronic post-surgical pain. The mechanism of action involves both peripheral and central actions. In addition to blockade of the Voltage-gated Sodium Channel of the peripheral nerves, lidocaine also inhibits priming of the PolyMorphoNuclear granulocyte (PMN) by inducing a time-dependent inhibition of intracellular G-protein signalling molecule (Gq); thus reducing release of cytokines and Reactive Oxygen Species Centrally, lidocaine also causes blockade of NMDA receptors and Neurokinin Receptors of the Wide-Dynamic Range Neurons in the dorsal horn of spinal cord; thus reduces glutamate activity.

We therefore hypothesize that the use of intravenous lidocaine may reduce acute pain and improve the range of knee ﬂexion after total knee replacement. Currently, there is strong evidence supporting its use in laparoscopic and open abdominal surgeries. There is, however, a paucity of studies in orthopedic surgeries. To date, there is no randomized controlled trial that studied its eﬀect in total knee replacement.

DETAILED DESCRIPTION:
OBJECTIVE:

The aim of this study is to estimate the effectiveness of a preemptive bolus of intravenous lidocaine on reduction in acute pain, improvement on the range of movement, other rehabilitation parameters and functional scoring in the post-operative period after total knee replacement.

DESIGN:

This is a double-blinded, randomized, placebo-controlled trial.

RECRUITMENT & SAMPLE SIZE:

Over a one-year period, suitable patients will be approached at the pre-admission clinic and in the general ward before their operation. Informed consent will be obtained before enrollment.

The sample size required is calculated to be 45 subjects per group.

PATIENT CHARACTERISTICS:

In order to minimize potential confounding factors, the demographic data of each subject will be collected during preoperative assessment, including: age, gender, duration of preoperative pain duration, preoperative NRS (movement) and NRS (rest). Both active and passive ROM of the knee will be assessed by the attending physiotherapist.

RANDOMIZATION & BLINDING:

Each subject will be assigned to either Lidocaine Group or Placebo Group. A randomization list will be established by a computer-generated random sequence before the study begins. An envelope containing the group assignment will be prepared, sealed, sequentially numbered, and allocated for each subject. A "blinded" anaesthetist will then prepare lidocaine or saline according to the group assigned for the attending anaesthetist. The subjects, the investigators, and all the parties involved in patient management or data collection will be blinded throughout the study period.

INTERVENTION:

For Lidocaine Group: a bolus of intravenous lidocaine of 2mg/kg over 5 mins will be given before skin incision.

For Placebo Group: Normal Saline of equal volume will be given as bolus before skin incision.

ANAESTHESIA & ANALGESIA:

(I) PRE-OPERATIVE: Routine preoperative assessment will be taken at the pre-admission clinic or at the general ward; and standard fasting times (6 hours for solid food and 2 hours for clear liquid) will be ordered.

No analgesics or sedatives will be given as pre-medication. Holter machine will be used to document any arrhythmia preoperatively and will be attached to patient till Day 1 postoperatively.

(II) INTRA-OPERATIVE: In addition to continuous ECG monitoring, BP, heart rate and SpO2 will be monitored at no longer than every 5 mins throughout the operation. Signs and symptoms of local anaesthetic toxicity will be assessed at 30 minute intervals.

After establishing at least one patent intravenous cannula and ensuring the monitors are properly applied, Spinal Anaesthesia will be given by the attending anaesthetist under aseptic technique.

The choice of equipment (Whitacre or Quincke Needle), technique (landmark or ultrasound-guided), and approach (midline or paramedical) are at the discretion of the attending anaesthetist.

An intrathecal dose of 2.2-2.6ml 0.5% Heavy Bupivacaine with 15mcg of fentanyl will be given depending on the height of the patient. Vasopressors and intravenous ﬂuids will be given as necessary to keep the patient's blood pressure within 20% of his/her baseline, and to keep the heart rate within normal range.

Bolus of lidocaine or placebo will then be given over 5 minutes before skin incision.

No Sedation will be given during operation in order to facilitate monitoring of systemic toxicity.

No Systemic Analgesics will be given, including Paracetamol, NSAIDS, Ketamine and Opioids.

The surgeries will be performed by the same team of orthopedic surgeons experienced in total knee replacement at a tertiary level university teaching hospital, using standardized surgical techniques. All patients will undergo posterior stabilized knee prosthesis.

Standardized dose of LIA (40ml 0.75% Ropivacaine, 0.5ml 1 in 200,000 Adrenaline, 30mg Ketorolac in 60ml Normal Saline) will be administered by the orthopedic team.

(III) POST-OPERATIVE (PHASE I RECOVERY IN PACU): Upon completion of surgery, the patient will be transferred to PACU for further monitoring for at least 30 minutes. BP, heart rate, and SpO2 will be monitored every 5 minutes in addition to continuous ECG monitoring. Signs and symptoms of local anaesthetic toxicity will be assessed at 15 minute intervals.

Pain will be evaluated every 5 mins using NRS. If the score is greater than 4/10, 2mg morphine will be given intravenously every 5 mins provided the patient has a respiratory rate of > 12/min and a sedation score of <1 until a NRS of < 4/10 is achieved. At which point, a patient-controlled analgesia (PCA) device will be connected to deliver morphine under a standardized regime: 1mg bolus with 5 mins lockout, an hourly maximum of 0.1mg/kg, and no background infusion.

(IV) POST-OPERATIVE (PHASE II RECOVERY IN WARD): Continuous ECG monitoring will continually be applied until Day 1 postoperatively.

Signs and symptoms of local anaesthetic toxicity will be assessed clinically at 1-hour intervals for 12 hours after operation.

BP, heart rate, SpO2, and sedation score will be monitored at 1-hour intervals while on PCA morphine; BP and heart rate will be monitored at 4-hour intervals once PCA morphine is terminated.

Postoperative analgesics will consist of:

PCA Morphine for at least 2 days postoperatively, and will be terminated on postoperative Day 3 once NRS (movement) is less than 4/10 or when 24-hour morphine consumption is less than 10mg.

Standardized analgesic regime, depending on body weight, will be started immediately after operation. For body weight > 50kg, Oral paracetamol 1gram QID, and pregabalin 75mg nocte for 1 week celecoxib 200mg BD for 5 days. For body weight < 50kg, Oral paracetamol 1gram TDS, and pregabalin 50mg nocte for 1 week. celecoxib 200mg daily for 5 days.

0.1mg/kg of intramuscular Morphine will be provided as necessary as rescue analgesic for any breakthrough pain. Intravenous Ondansetron of 0.1mg/kg will be given as necessary for nausea and vomiting.

Diet will be resumed on Postoperative Day 0. The rehabilitation programme will be standardized for all patients and be carried out by the same team of physiotherapists and occupational therapists with the goal of early mobilization on Postoperative Day 0.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Primary Elective Total Knee Replacement under Spinal Anaesthesia

Exclusion Criteria:

* Single Stage Bilateral Total Knee Replacement
* Revision Total Knee Replacement
* Contraindications to Spinal Anaesthesia or Failed Spinal Anaesthesia
* Allergy to amide local anaesthetics, paracetamol, non-steroidal anti-inflammatory drugs (NSAIDS), opioids
* Cardiac Disease: Any degree of Heart Block, Heart Failure
* Neurological: Any Seizure Disorder
* Psychiatric illnesses affecting pain perception e.g. severe depression and anxiety disorder
* Alcohol or substance abuse
* Chronic Pain, other than chronic knee pain
* Daily use of strong opioids (morphine, fentanyl, hydromorphone, ketobemidone, methadone, nicomorphine, oxycodone, or meperidine)
* Impaired Renal Function (defined as preoperative serum creatinine level over 200µmol/L)
* Impaired Hepatic Function
* Pregnancy
* Inability to use PCA
* Patient Refusal
* Patients do not understand Cantonese

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
Pain assessed by numerical rating scales (NRS) pain scores | at postoperative day 1
  NRS pain scores (from 0-10, where 0 is the least satisfaction and 10 most satisfaction) will be recorded during movement and at rest, by NRS (movement) and NRS (rest) respectively

SECONDARY OUTCOMES:
Range of motion (ROM) of knee | until postoperative day 6
  Active and Passive ROM of knee (flexion and extension) will be recorded.
Availability of usual activity of knee | until postoperative day 6
  Walking Distance, degree of assistance, and need for aids
Self Care Assessment | until postoperative day 6
  Dressing trousers, toileting will be recorded
Side Effects of PCA Morphine | until postoperative day 6
  Nausea, vomiting, dizziness, constipation

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong